CLINICAL TRIAL: NCT05015699
Title: A Prospective, Multi-center, Single-group Target Value Post-marketing Clinical Study to Evaluate the Safety and Effectiveness of the HT Supreme Drug-eluting Stent System in the Treatment of "Real-world" Patients With Coronary Heart Disease
Brief Title: A Study to Evaluate the Impact of 11-month Ticagrelor Monotherapy Following One-month DAPT After PCI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawn of the research project based on the company's decision
Sponsor: Sino Medical Sciences Technology Inc. (Industry)
Collaborators: The Second Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PIONEER IV CHINA
Record Dates: First submitted 2021-08-01; First posted 2021-08-20 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Coronary Artery Disease
Keywords: Healing-Targeted Supreme; one month DAPT
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HT Supreme (Experimental): Device: HT Supreme ( R&D by Sinomed, Tianjin, China) Drug: 11-month ticagrelor monotherapy following one-month dual antiplatelet therapy (DAPT) after HT Supreme drug-eluting stent system interventions
  Interventions: Device: HT Supreme

INTERVENTIONS:
Device: HT Supreme — HT Supreme ( R&D by Sinomed, Tianjin, China)

SUMMARY:
PIONEER IV CHINA is sought to investigate the safety and efficacy of 11-month ticagrelor monotherapy following one-month dual antiplatelet therapy (DAPT) after HT Supreme drug-eluting stent system at 12 months follow-up.

DETAILED DESCRIPTION:
This study is a prospective, multi-center, single-arm objective performance criteria clinical trial in an all-comers patient population (including patients with high bleeding risk, HBR) undergoing PCI with unrestrictive use of the HT Supreme sirolimus-eluting stent and treated with 11-month ticagrelor monotherapy following one-month dual antiplatelet therapy (DAPT) in approximately 285 patients (including 80 coronary heart disease cases entering the OCT subgroup). All patients will be (at minimum) contacted via visit at 30 days (±7 days) and at 12 months (±30 days), and by phone contact at 6 months (±14 days), 24 months (±30 days) and 36 months (±45 days) post index procedure to assess clinical status and adverse events. The Primary Endpoint for this trial is Patient-oriented Composite Endpoint (PoCE) at 12 months post-procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient ≥18 years of age;
2. Patient has chronic stable angina, acute coronary syndromes or silent ischemia;
3. Presence of one or more coronary artery stenoses of ≥50% (by visual assessment) in a native coronary artery (with or without prior stent/other device treatment) or in a saphenous venous or arterial bypass conduit suitable for coronary stent implantation;
4. The vessel should have a reference vessel diameter of at least 2.25 mm by visual assessment (no limitation on the number of treated lesions, vessels, or lesion length);
5. Patient has been informed of the nature of the study and agrees to its provisions and has provided written informed consent as approved by the Ethical Committee and is willing to comply with all protocol-required (follow-up) evaluations.

Exclusion Criteria:

1. under 18 years of age;
2. Unable to sign written informed consent
3. Patient is a woman who is pregnant or nursing
4. Known intolerance to cobalt chromium, and medications such as sirolimus, aspirin, heparin, bivalirudin or P2Y12 inhibitors;
5. Planned major elective surgery requiring discontinuation of DAPT within 12 months of procedure;
6. Concurrent medical condition with a life expectancy of less than 3 years;
7. Currently participating in another trial and not yet at its primary endpoint
8. Active pathological bleeding;
9. History of intracranial haemorrhage.

OCT exclusion criteria

1. Left main lesion
2. Severe tortuous, calcified or angulated coronary anatomy of the study vessel that in the opinion of the investigator would result in suboptimal imaging or excessive risk of complication from placement of an OCT catheter
3. Total occlusion or thrombolysis in myocardial infarction(TIMI) flow 0, prior to wire crossing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Rate of Patient-oriented Composite Endpoint (PoCE) at 12 months post-procedure. | 12 months post-procedure
  PoCE is a composite clinical endpoint of: all-cause death; any stroke, Modified Rankin scale, (MRS ≥1); any myocardial infarction (peri-procedural MI according to SCAI, spontaneous according to 4th universal definition); any clinically and physiologically driven revascularization (ARC-2)

SECONDARY OUTCOMES:
Rate of Patient oriented composite endpoint (PoCE) at 2 and 3 years; | 2 and 3 years post-procedure
  PoCE is a composite clinical endpoint of: all-cause death; any stroke, Modified Rankin scale, (MRS ≥1); any myocardial infarction (periprocedural MI according to SCAI, spontaneous according to 4th universal definition); any clinically and physiologically driven revascularization (ARC-2)
Rate of Individual components of patient-oriented composite endpoint; | 1, 2 and 3 years post-procedure
  PoCE is a composite clinical endpoint of: all-cause death; any stroke, Modified Rankin scale, (MRS ≥1); any myocardial infarction (periprocedural MI according to SCAI, spontaneous according to 4th universal definition); any clinically and physiologically driven revascularization (ARC-2)
Rate of Vessel-oriented composite endpoints (VoCE) | 1, 2 and 3 years post-procedure
  VoCE is a composite clinical endpoint of: Vessel-related cardiovascular Death; Target-vessel related MI; Clinically and physiologically-oriented Target vessel revascularization (ARC-2)
Rate of Individual components of vessel-oriented composite endpoint; | 1, 2 and 3 years post-procedure
  VoCE is a composite clinical endpoint of: Vessel-related cardiovascular Death; Target-vessel related MI; Clinically and physiologically-oriented Target vessel revascularization (ARC-2)
Rate of Device-oriented composite endpoint (DoCE) at all timepoints; | 30days, 6months, annually up to 3 years post procedure
  VoCE is a composite clinical endpoint of: Cardiovascular Death；Target-vessel related MI；Clinically and physiologically-oriented Target lesion revascularization
Rate of Individual components of device-oriented composite endpoint; | 30days, 6months, annually up to 3 years post procedure
  VoCE is a composite clinical endpoint of: Cardiovascular Death；Target-vessel related MI；Clinically and physiologically-oriented Target lesion revascularization
Rate of Pre-procedural myocardioal infarction according to 4th universal definition; | 30days, 6months, annually up to 3 years post procedure
  Fourth Universal Definition of Myocardial Infarction (2018)
Device Success Rate | intra-operative
  according to the statement from European Association of Percutaneous Cardiovascular Interventions (EAPCI) of the European Society of Cardiology (ESC))
Rate of Stent thrombosis | 30days, 6months, annually up to 3 years post procedure
  Stent thrombosis is consist of Definite stent thrombosis; Probable stent thrombosis; Definite or probable stent thrombosis
Rate of Target-vessel failure composite endpoint | 30days, 6months, annually up to 3 years post procedure
  TVF is a composite clinical endpoint of: Cardiac death; Myocardial Infarction (MI) (unless clearly attributable to a non target vessel); Target vessel revascularization
Rate of Individual components of Target-vessel failure composite endpoint | 30days, 6months, annually up to 3 years post procedure
  TVF is a composite clinical endpoint of: Cardiac death; Myocardial Infarction (MI) (unless clearly attributable to a non target vessel); Target vessel revascularization
Rate of Bleeding according to BARC (2, 3 and 5) classification | 30days, 6months, annually up to 3 years post procedure
  Defining high bleeding risk in patients undergoing percutaneous coronary intervention: a consensus document from the Academic Research Consortium for High Bleeding Risk
Rate of Net adverse clinical and cerebral events | 30days, 6months, annually up to 3 years post procedure
  NACCE is a composite clinical endpoint of: any cause, myocardial infarction (MI), cerebral vascular accident, and major bleeding (according to the modified REPLACE-2 and GUSTO criteria)
Cost-Effectiveness | hospitalization, 1 year post procedure
  Cost of procedure will be collected in the eCRF(e.g. diagnostic tests, procedural materials, time of the procedure, re-angiography, repeat revascularization, etc. will be quantified).

OTHER OUTCOMES:
The percentage of the struts' neointimal coverage (%) measured by OCT | 1 month post procedure
  80 patients enrolled with an extra one-month OCT follow-up as a subgroup analysis target. OCT examination was carried out at 1 month after the operation to evaluate percentage of the struts' neointimal coverage
Neointimal hyperplasia area/volume measured by OCT | 1 month post procedure
  80 patients enrolled with an extra one-month OCT follow-up as a subgroup analysis target. OCT measures Neointimal hyperplasia area(mm2)/volume(mm3)
Mean/Minimal Stent diameter/area/volume | 1 month post procedure
  80 patients enrolled with an extra one-month OCT follow-up as a subgroup analysis target. OCT measures Mean/Minimal Stent diameter(mm)/area(mm2)/volume(mm3)
Mean/maximal thickness of the struts coverage(%) | 1 month post procedure
  80 patients enrolled with an extra one-month OCT follow-up as a subgroup analysis target. OCT measures Mean/maximal thickness of the struts coverage
Mean/Minimal Lumen diameter/area/volume | 1 month post procedure
  80 patients enrolled with an extra one-month OCT follow-up as a subgroup analysis target. OCT measures Mean/Minimal Lumen diameter(mm)/area(mm2)/volume(mm3)
Incomplete strut apposition（%） | 1 month post procedure
  80 patients enrolled with an extra one-month OCT follow-up as a subgroup analysis target. OCT examination was carried out at 1 month after the operation to evaluate incomplete strut apposition

CONTACTS AND LOCATIONS:
Overall Officials: Bo Yu, PH.D, Principal Investigator — The Second Affiliated Hospital of Harbin Medical University; Haibo Jia, PH.D, Study Director — The Second Affiliated Hospital of Harbin Medical University